CLINICAL TRIAL: NCT06342895
Title: Interpretation and Optimization of Nutrition in the Intensive Care Units
Acronym: IONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dim3 (Industry)
Collaborators: Baxter Healthcare Corporation (Industry); University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020_1113; 2022-A00103-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Nutritional Support
Keywords: Intensive Care Unit; Protein Calorie Malnutrition; Refeeding syndrome; Clinical Decision Support Systems
MeSH Terms: conditions — Protein-Energy Malnutrition; Refeeding Syndrome

STUDY DESIGN:
Intervention Model Description: Usual use of standard clinical and biological information related to nutritional support as available through the ICU electronic health record (i.e. without any calculated information on recommended, prescribed, or received calories and protein, only information on prescribed products and volumes as collected by and presented in the ICU EHR) In this arm, participants, investigators, and healthcare professionals will be blinded to real-time enteral feed volumes that will be collected by the Feedim medical device and transmitted to the electronic study case report form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental)
  Interventions: Device: Nutritional support prescription and delivery monitoring feedback
- control (Other)
  Interventions: Device: Usual care

INTERVENTIONS:
Device: Nutritional support prescription and delivery monitoring feedback — Real-time availability in an integrated computer interface (Nutrow) of all clinical and biological information related to nutritional support including recommended, prescribed, and delivered calories and proteins and enteral feed delivery transmitted by the Feedim medical device
  Arms: Interventional
Device: Usual care — Usual use of standard clinical and biological information related to nutritional support as available through the ICU electronic health record (i.e. without any calculated information on recommended, prescribed, or received calories and protein, only information on prescribed products and volumes as collected by and presented in the ICU EHR) In this arm, participants, investigators, and healthcare professionals will be blinded to real-time enteral feed volumes that will be collected by the Feedim medical device and transmitted to the electronic study case report form.
  Arms: control

SUMMARY:
Despite recommendations, inadequate nutritional intake in intensive care unit (ICU) patients remains frequent and can lead to complications such as infections, increased length of stay, prolonged weaning from ventilation, increased long-term mortality, and decreased quality of life after intensive care. Studies have shown that patients only receive up to 50-60% of prescribed calories and proteins due to many factors leading to nutritional support interruptions such as ICU procedures, physical therapy, transport for imaging or invasive procedures outside the ICU, and nutrition intolerance.

Furthermore, this discrepancy between prescribed and delivered nutrition may go largely unnoticed, due to issues concerning inadequate manual or automated monitoring of delivered nutrition. A joint "Call to Action" by ASPEN, the Academy of Nutrition and Dietetics, and the American Society of Health-System Pharmacists stated that parenteral nutrition errors and their contributing factors could be prevented by improving the functionality of in-house Clinical Decision Support Systems and the interfaces between electronic health records (EHRs), automated preparation devices and pharmacy systems.

Nutrow® is a software package designed to support nutritional management based on the calculation of recommended calorie and protein requirements, real-time calculation and monitoring of calorie and protein prescriptions, real-time calculation and monitoring of calories and protein truly delivered to patients, and information feedback to prescribers. Feedim® is a Medical Device Data System (MDDS), designed by Dim3, which transmits information from enteral feeding pumps to third-party software, such as Nutrow®.

The aim of the study is to assess whether the joint use of Nutrow-Feedim improves the achievement of nutritional objectives in ICU patients prior to oral intake by reducing the discrepancy between prescribed and delivered calories and protein.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over.
* French Social Security system registration.
* First stay in ICU
* Admitted to the Lille University Hospital Surgical ICU for at least 3 days.
* Active enteral and/or parenteral nutritional support prescription
* Patient and/or next-of-kin informed about the study and having consented to participation in the study.

Exclusion Criteria:

* Age under 18
* Burn patient
* Admitted to the ICU with a prior active enteral/parenteral nutritional support before day 3, except trophic nutrition
* Dying patient, not-to-be-resuscitated order, or other treatment limitation decision at ICU admission
* Adult under guardianship
* Department of corrections inmate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Mean total daily calories delivered/prescribed ratio (percent) | From ICU Day 3 to Day 28 or until any of the following if before day 28: Return to oral intake Discharge from the ICU Death
  Total (enteral+parenteral) prescribed and delivered calories are measured daily (kcal/day).
  The ratio of mean total daily delivered calories over the study period divided by the mean total daily prescribed calories over the study period will be calculated and expressed as a %

SECONDARY OUTCOMES:
Mean total daily protein delivered/prescribed ratio (%) | From ICU Day 3 to Day 28 or until any of the following if before day 28: Return to oral intake Discharge from the ICU Death
  Total (enteral+parenteral) prescribed and delivered protein are measured daily (g/day).
  The ratio of total mean daily delivered protein over the study period divided by the mean total daily prescribed protein over the study period will be calculated and expressed as a %
Mean total daily calories delivered/recommended ratio (percent) | From ICU Day 3 to Day 28 or until any of the following if before day 28: Return to oral intake Discharge from the ICU Death
  Total (enteral+parenteral) prescribed and delivered calories are measured daily (kcal/day).
  The ratio of mean total daily delivered calories over the study period divided by the mean total daily recommended calories (according to guidelines) over the study period will be calculated and expressed as a %
Mean total daily protein delivered/recommended ratio (percent) | From ICU Day 3 to Day 28 or until any of the following if before day 28: Return to oral intake Discharge from the ICU Death
  Total (enteral+parenteral) prescribed and delivered protein are measured daily (g/day).
  The ratio of mean total daily delivered protein over the study period divided by the mean total daily recommended protein (according to guidelines) over the study period will be calculated and expressed as a %
Nutritional support duration (days) | From ICU Day 3 to Day 28 or until any of the following if before day 28: Return to oral intake Discharge from the ICU Death
  Days on nutritional support (either parenteral and/or enteral) over the study period
Time to initiation of nutritional support (days) | From ICU Day 3 to Day 28 or until any of the following if before day 28: Return to oral intake Discharge from the ICU Death
  Days elapsed from ICU admission (Day 1) to first administration of any nutritional support (either parenteral and/or enteral) over the study period
Weight (Kg) | From ICU Day 3 to Day 28 or until any of the following if before day 28: Return to oral intake Discharge from the ICU Death
  Daily body weight (Kg) as weighed using weighing scale integrated in the ICU-bed
Day 28 mortality rate | From ICU admission (Day1) to Day 28
  Patient death during the timeframe
ICU length-of-stay (days) | From ICU admission (Day1) to ICU discharge, data censored at Day 28 max
  Days patient present in the ICU
Days on ventilator (days) | From ICU admission (Day1) to ICU discharge, data censored at Day 28 max
  Days patient on ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Eric KIPNIS, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided